CLINICAL TRIAL: NCT04752852
Title: Randomised Control Trial on the Use of Prophylactic Steroids in the Prevention of Post-thyroidectomy Hypocalcaemia and Voice Dysfunction
Brief Title: Use of Prophylactic Steroids in the Prevention of Post-thyroidectomy Hypocalcaemia and Voice Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holy Family Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Raheel Ahmad, Principal Investigator, Holy Family Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 233/HFH12/14
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Thyroid Diseases; Hypocalcemia; Vocal Cord Dysfunction
Keywords: Thyroidectomy; Postoperative Hypocalcaemia; Postoperative Vocal cord dysfunction; Dexamethasone
MeSH Terms: conditions — Thyroid Diseases; Hypocalcemia; Vocal Cord Dysfunction | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Patients with odd numbers were assigned to group A. 8 mg/2 ml dexamethasone was injected intravenously sixty minutes before the induction of anaesthesia
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Patients with even numbers were assigned to group B. Two millilitres (ml) normal saline (0.9%) was given intravenously 60 minutes before the induction of anaesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 8 mg/2 ml dexamethasone IV, 60 minutes before the induction of anaesthesia
  Arms: Dexamethasone
Drug: Placebo — 2 ml normal saline (0.9%) IV, 60 minutes before the induction of anaesthesia
  Other Names: normal saline (0.9%)
  Arms: Placebo

SUMMARY:
Total thyroidectomy for benign surgical pathologies is associated with risks related to temporary hypocalcaemia and vocal quality dysfunction. Dexamethasone, as an anti-inflammatory steroid, has been proposed to have a physiological effect on hypocalcaemia and voice quality. Investigators conducted a double-blinded controlled trial to assess the effect of preoperative dexamethasone on the vocal dysfunction and hypocalcaemia following thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* Benign thyroid condition.
* Patients without any preoperative corrected hypocalcaemia and voice or vocal quality dysfunction.

Exclusion Criteria:

* Previous thyroid or neck surgery
* Known vocal cord dysfunction on laryngoscopy
* Hearing or voice problems
* History of gastroesophageal reflux and stomach ulcer disease
* Contraindications of steroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Hypocalcaemia | 3 days
  Hypocalcaemia was defined as a corrected serum calcium level of less than 2 mmol/L.
Voice dysfunction | 24 hours
  Signs and symptoms of voice dysfunction at 24 hours after thyroidectomy. Voice dysfunction was defined on voice analogue score from 0-100. Participants with Voice Analogue Score of less than 50 were labelled as having voice dysfunction, and participants with score more than 50 were considered as normal.

CONTACTS AND LOCATIONS:
Overall Officials: Raheel Ahmad, FCPS, Principal Investigator — Holy Family Hospital Rawalpindi Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Worni M, Schudel HH, Seifert E, Inglin R, Hagemann M, Vorburger SA, Candinas D. Randomized controlled trial on single dose steroid before thyroidectomy for benign disease to improve postoperative nausea, pain, and vocal function. Ann Surg. 2008 Dec;248(6):1060-6. doi: 10.1097/SLA.0b013e31818c709a. PMID 19092351
- [Background] Kolahdouzan M, Iraj B, Eslamian M, Harandizadeh M, Meamar R. Preventive Effect of Dexamethasone Therapy on the Transient Hypoparathyroidism through Total Thyroidectomy. Iran J Otorhinolaryngol. 2019 Mar;31(103):73-80. PMID 30989072
- [Derived] Dhahri AA, Ahmad R, Rao A, Bhatti D, Ahmad SH, Ghufran S, Kirmani N. Use of Prophylactic Steroids to Prevent Hypocalcemia and Voice Dysfunction in Patients Undergoing Thyroidectomy: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Oct 1;147(10):866-870. doi: 10.1001/jamaoto.2021.2190. PMID 34473215